CLINICAL TRIAL: NCT04633109
Title: The Obese Taste Bud Study
Acronym: OTB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Collaborators: Helmholtz Institut für Metabolismus-, Adipositas- und Gefäßforschung (Unknown); Klinik und Poliklinik für Hals-, Nasen- und Ohrenheilkunde (Unknown); Klinik und Poliklinik für Mund-, Kiefer- und Plastische Gesichtschirurgie (Unknown); Poliklinik für Zahnärztliche Prothetik und Werkstoffkunde (Unknown)
Responsible Party: Principal Investigator, Imke Schamarek, Clinician Scientist, University of Leipzig
Other Study IDs: OTB-2020; DRKS00022950 (Registry Identifier: DRKS)
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Obesity; food preferences; taste disorder; taste bud; metabolic disease; feeding behavior
MeSH Terms: conditions — Obesity; Food Preferences; Taste Disorders; Metabolic Diseases; Feeding Behavior | interventions — Glucose Tolerance Test; Anthropometry; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Taste buds, saliva, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal weight: Normal weight adults with BMI ranging from 18.5-24.9; men and women; age range 18-69years; written informed consent
  Interventions: Procedure: taste bud biopsy; Diagnostic Test: oral glucose tolerance test; Diagnostic Test: Taste sensitivity; Diagnostic Test: olfactory function; Diagnostic Test: taste bud density; Diagnostic Test: anthropometry; Other: biospecimen collection; Other: questionnaires
- obese: Subjects with obesity as defined by BMI >= 30; men and women; age range 18-69 years; written informed consent
  Interventions: Procedure: taste bud biopsy; Diagnostic Test: oral glucose tolerance test; Diagnostic Test: Taste sensitivity; Diagnostic Test: olfactory function; Diagnostic Test: taste bud density; Diagnostic Test: anthropometry; Other: biospecimen collection; Other: questionnaires

INTERVENTIONS:
Procedure: taste bud biopsy — Taste buds will be surgically removed a) during a planned and medically induced elective surgery under full anesthesia; b) by local anesthesia in subjects without a medically induced surgery
Diagnostic Test: oral glucose tolerance test — 75g glucose will be applied in drinking water following blood sample collection to evaluate glucose, insulin and C-peptide level.
Diagnostic Test: Taste sensitivity — Subjects are given taste strips with 4 concentrations per each taste quality of sweet, sour, salty, bitter and umami in a pseudo-randomized manner. Subjects are asked to identify the taste quality, state the intensity, preference and certainty.
Diagnostic Test: olfactory function — Subjects will be presented 16 different sniffing sticks in a randomized order, each for about 4seconds. People are then asked to identify the smell by choosing one out of 4 options (forced choice).
Diagnostic Test: taste bud density — The number of taste buds on the anterior tongue will be determined by colouring the tongue surface with food colour. Taste buds will apply more reddish as compared to non-taste tissue. Based on a digital photography the number of taste buds per subjects is counted manually.
Diagnostic Test: anthropometry — Anthropometric data collection will include measures of body height, body weight, arm-, upper- and lower leg circumferences, waist- and hip circumferences and a bioimpedance analysis to obtain data about body composition.
Other: biospecimen collection — Blood and saliva samples will be taken as well as a tongue swab.
Other: questionnaires — Through the use of several questionnaires, data about eating behavior, food preferences, life style factors and other will be obtained.

SUMMARY:
The sense of taste is essential for priming food preferences and is therefore important for caloric uptake and body weight regulation. Recent studies show that obesity is linked to changes in taste sensation but also to a loss of taste buds on the tongue. This study aims to evaluate underlying mechanisms within the taste buds to potentially influence the sense of taste on the level of these sensory cells and in order to develop new treatment strategies to fight obesity.

ELIGIBILITY:
Inclusion Criteria:

* normal weight (BMI 18.5-24.9)
* obesity (BMI >=30)
* overall healthy (no severe sickness, no cancer)
* written informed consent

Exclusion Criteria:

* current pregnancy or currently breastfeeding
* cancer or tumors
* state after radiotherapy at head-neck area
* state after or current chemotherapy
* severe psychiatric-, cardiac-, kidney- or neurological illness
* diagnosed diabetes mellitus
* known dysfunction of smelling or tasting
* drug or alcohol abuse
* permanent medication with antidepressants, anticonvulsants, steroids and/or immunosuppressants

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study population will mainly consits of patients who underwent a medically induced elective surgery at the head or neck area (f.e. surgery at the soft palate, plastic surgery, maintenance of congenital anomalies etc.) or healthy participants recruited elsewhere at the campus area of the Medical Faculty of the University of Leipzig, Saxony, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Identification of differential gene and protein regulation in isolated human taste cells between lean and obese subjects | through study completion, an average of 2 years
  Transcriptomics (RNAsequencing (seq), single cell seq) and epigenomics (open chromatin mapping (ATACseq), Infinium MethylationEPIC Array) will be performed in isolated papillae fungiformes. Validation analyses by in vitro primary cell cultures of taste cell biopsy
Identification of correlations between taste cell biology with parameters of intervention | 1 year
  corrleation analyses will include factors of eating behavior, food preferences, life style factors, data from taste and smell screenings, anthropometric data, blood and saliva parameters

SECONDARY OUTCOMES:
Differences of salivary and tongue microbiome on taste cells in obesity in contrast to lean | 2 years
  whole mouth saliva as well as local tongue microbiome diversity will be analysed by 16S ribosomal RNA seq and related to further parameters of this study.
extracellular vesicle analyses of saliva in lean and obese subjects | 2 years
  The content of extracellular vesicles from saliva samples will be analysed and compared between the study groups as well as related to other parameters of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stumvoll, Prof. Dr., Study Director — Medical Faculty of the University of Leipzig, Leipzig, Germany; Imke Schamarek, Dr., Principal Investigator — Medical Faculty of the University of Leipzig, Leipzig, Germany
Locations (1):
- Medical Clinic III, Division of Endocrinology, University Clinic of Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
one aim of this study is to obtain large-scale sequencing data. with this several not yet defined research questions will be generated which shall be explored through later analyses and projects. in order to exploit the potential of the data and to avoid misinterpretation, the data should only be accessible to the scientists and collaborators involved.